CLINICAL TRIAL: NCT03101761
Title: Characteristics and the Future of the City Chilblains
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ENGELURES
Record Dates: First submitted 2017-03-17; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Chilblains
MeSH Terms: conditions — Chilblains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chilblains are cutaneous lesions affecting extremities (foot and fingers) with erythemic papules, evolving by painful relapse due to cold and sudden reheating.

This pathology is currently poorly understood while it's frequent.

The aim of the study is to evaluate all the characteristics of this pathology by reporting clinical and biological data of patient consulting for chilblains; and the other point is to assess the evolution of these patients.

DETAILED DESCRIPTION:
Investigators are going to collect data on patient medical report to fill up a case report form. And in a second time they call patient by phone to ask him/her about the evolution of their pathology.

ELIGIBILITY:
Inclusion Criteria:

* patient consulting for chilblains
* diagnostic of chilblain during the consultation

Exclusion Criteria:

* patients consulting for other reason than chilblains
* patient who can't reply by telephonic call

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient consulting for chilblains between 2012 and 2014
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Évaluation of chilblains' topography | Day 1
  This assessment consists to evaluate the chilblains topography, vasospastic profile and presence or not of another acrosyndrome

SECONDARY OUTCOMES:
Questionnaire of assessment of chilblains' evolution | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PRIOLLET, MD, Study Director — Groupe Hospitalier Paries St JOSEPH
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No